CLINICAL TRIAL: NCT04911881
Title: A Phase Ia, Open-Label, Multi-Center, Study of the Safety, Tolerability and Primary Efficacy of IBI321 in Patients With Advanced Solid Tumors
Brief Title: A Study of the Safety and Tolerability of IBI321 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI321A101
Record Dates: First submitted 2021-05-25; First posted 2021-06-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ia Dose-Escalation Stage: IBI321 (Experimental)
  Interventions: Drug: IBI321

INTERVENTIONS:
Drug: IBI321 — Several dose levels will be evaluated for IBI321 administered as a single agent. IBI321 will be given via IV infusion on Day 1 of each cycle until disease progression or loss of clinical benefit.

SUMMARY:
This first-in-human open-label,dose-escalation study is designed to evaluate the safety, tolerability, and primary efficacy of IBI321 in participants with locally advanced, recurrent, or metastatic incurable tumors for whom standard therapy does not exist, has proven to be ineffective or intolerable.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to give voluntary informed consent, understand the study and are willing to follow and complete all the test procedures.
2. Patients with advanced solid tumors who had failed standard treatment.
3. Male or female subjects ≥18 years and ≤75 years.
4. At least one measurable lesion per RECIST version 1.1
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
6. Life expectancy of ≥ 12 weeks.
7. Adequate hematologic and end organ function

Exclusion Criteria:

1. Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, targeted therapy, or immunotherapy.
2. Failure to recover from adverse events from the most recent anti-tumor treatment
3. Acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
4. Subjects with CNS metastasis unless they are asymptomatic or adequately treated with radiotherapy and/or surgery and subjects are neurologically stable with minimal residual symptoms/signs.
5. Any other serious underlying medical (e.g., uncontrolled hypertension, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, other serious cardiac conditions not listed in exclusion criteria), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.
6. Pregnancy, lactation, breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | From Day 1 of Cycle 1 to Day 28
Percentage of Participants with Adverse Events (AEs), treatment-related AE (TRAE), immune-related AEs (irAE) and serious adverse event (SAE) per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 ; | From Day 1 to up to 2 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR)per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. | From Baseline until disease progression (up to 2 years)
Progression Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. | From Baseline until disease progression (up to 2 years)
Duration of Response (DoR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. | From Baseline until disease progression (up to 2 years)
Overall Survival (OS) | From Baseline until disease progression (up to 2 years)
Area Under the Concentration-Time Curve (AUC) of IBI321 | From Day 1 up to 2 years
Maximum Serum Concentration (Cmax) of IBI321 | From Day 1 up to 2 years
Minimum Serum Concentration (Cmin) of IBI321 | From Day 1 up to 2 years
Clearance (CL) of IBI321 | From Day 1 up to 2 years
Percentage of Participants with Anti-Drug Antibodies (ADAs) and Neutralizing Antibody (Nab) to IBI321 | From Day 1 up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China